CLINICAL TRIAL: NCT05632328
Title: A Phase 2 Study of AGEN1423, an Anti-CD73-TGFβ-Trap Bifunctional Antibody, in Combination With Botensilimab, With or Without Chemotherapy in Subjects With Advanced Pancreatic Cancer.
Brief Title: AGEN1423 and Botensilimab w/ or w/o Chemo in PDAC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bruno Bockorny (Other)
Collaborators: Agenus Inc. (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Bruno Bockorny, Principal Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-213
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Advanced Pancreatic Ductal Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: Advanced Pancreatic Ductal Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Chemotherapy; Immunotherapy; AGEN1423; Botensilimab
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- COHORT 1: AGEN1423 Plus Botensilimab (Experimental): Treatment is AGEN1423 plus Botensilimab for 4 cycles (8 weeks) followed by Botensilimab alone for up to 2 years. AGEN1423 will be administered in a total of 4 doses. Botensilimab will be administered every 2 weeks.
  Interventions: Drug: AGEN1423; Drug: Botensilimab
- COHORT 2: AGEN1423 Plus Botensilimab and Chemotherapy (Experimental): Treatment is AGEN1423 plus Botensilimab in combination with gemcitabine and nab-paclitaxel for 2 cycles (8 weeks) followed by Botensilimab in combination with gemcitabine and nab-paclitaxel for up to 2 years. AGEN1423 will be administered in a total of 4 doses. Botensilimab will be administered once every 2 weeks.
  Interventions: Drug: AGEN1423; Drug: Botensilimab; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: AGEN1423 — via IV, dosage per protocol, once every 2 weeks for up to 8 weeks
  Other Names: Anti-CD73-TGFβ-Trap Bifunctional Antibody
Drug: Botensilimab — via IV, dosage per protocol, once evert 2 weeks, up to 2 years
Drug: Gemcitabine — per standard care
  Other Names: Gemzar
  Arms: COHORT 2: AGEN1423 Plus Botensilimab and Chemotherapy
Drug: Nab-paclitaxel — per standard care
  Other Names: Abraxane
  Arms: COHORT 2: AGEN1423 Plus Botensilimab and Chemotherapy

SUMMARY:
The goal of this research study is to asses the safety and efficacy of the combination of AGEN1423 and Botensilimab with or without chemotherapies, gemcitabine and nab-paclitaxel, for the treatment of advanced pancreatic ductal adenocarcinoma (PDAC) which has progressed after at least one previous line of cancer therapy.

The names of the study drugs involved in this study are:

* AGEN1423
* Botensilimab

Participants will receive study treatment for about 2 years and will be followed for 1 year after.

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* Participants will receive study treatment for about 2 years and will be followed for 1 year. If the combination is considered to be safe and tolerable, and objective response is achieved in at least 2 patients, the study will proceed to Cohort 2.
* This research study involves immunotherapy. The names of the study drugs involved in this study are:
* AGEN1423
* Botensilimab

It is expected that about 24 people will take part in this part of this research

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved AGEN1423 as a treatment for any disease. The U.S. Food and Drug Administration (FDA) has not approved Botensilimab as a treatment for any disease.

Agenus, a pharmaceutical company, is supporting this research study by providing funding and study drug for the research study.

ELIGIBILITY:
Inclusion Criteria:

* 18 year and older
* Ability to understand and willingness to sign a written informed consent prior to entering the study.
* Histologically or cytologically confirmed (either previously or newly biopsied) metastatic or locally advanced unresectable pancreatic adenocarcinoma, including intraductal papillary mucinous neoplasm.
* Have measurable disease (≥ 1 measurable lesion) based on RECIST v1.1 as determined by the site study team. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Previous treatment lines

  * Cohort 1: Have documented objective radiographic progression on or after stopping treatment with first-line or further therapy, i.e. chemotherapy and or radiotherapy. If subjects received prior neoadjuvant or adjuvant chemotherapy and progressed within 3 months of the last dose, then this should be considered as a prior line of systemic therapy.
  * Cohort 2: Have documented objective radiographic progression on or after stopping treatment with first-line, fluorouracil-based chemotherapy.
* For Cohort 1, willing to submit an evaluable fresh tumor tissue sample, unless tumor is considered inaccessible, or biopsy is otherwise considered not in the subject's best interest.
* Complete resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia and peripheral neuropathy). If the subject received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
* ECOG status ≤1
* Life expectancy of at least 3 months
* Participants must have adequate organ and marrow function as defined below. All laboratory assessments should be performed within 10 days of treatment initiation

  * Hematological:

    * Hemoglobin ≥ 9g/dL (without transfusion within 7 days of assessment)
    * Leukocytes ≥3,000/µL
    * Absolute neutrophil count ≥1,500/µL
    * Absolute lymphocyte count ≥700/µL
    * Platelets ≥100,000/µL
  * Hepatic Function

    * Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * Renal Function

    ---Creatinine Clearance > 50 mL/min as calculated per Cockcroft-Gault formula
  * Nutritional

    ---Serum Albumin ≥ 3 g/dL
  * Coagulation

    * INR or PT: ≤1.5xULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
    * aPTT: ≤1.5xULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Subjects must use effective contraception:

  * Female subjects must be of non-childbearing potential or, if of childbearing potential, must agree to use a highly effective method of birth control (Appendix B), during the study and for 6 months following the last dose of study medication and must have a negative urine or serum pregnancy test within 72 hours prior to taking study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible. Non-childbearing potential is defined as (by other than medical reasons):

    ---≥45 years of age and has not had menses for over 2 years

    ---Amenorrhoeic for > 2 years without a hysterectomy and oophorectomy
  * Post hysterectomy, bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation at least 6 weeks prior to Screening. Information must be captured appropriately within the medical records.
  * Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Has a pancreatic tumor other than adenocarcinoma, including: adenosquamous, acinar cell carcinoma, pancreaticoblastoma, malignant cystic neoplasms, endocrine neoplasms, squamous cell carcinoma, Vater and periampullary duodenal or common bile duct malignancies.
* Subjects with a bowel obstruction.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has an active infection requiring systemic therapy or has an uncontrolled infection.
* Has an underlying medical condition that would preclude study participation.
* Has a disease that is suitable for therapy administered with curative intent.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from AE due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at Baseline) from AE due to a previously administered agent (Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study. If subject underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy)
* An active autoimmune disease that has required systemic treatment in the 2 years preceding the study (i.e., with the use of disease-modifying agents, corticosteroids or immuno-suppressive drugs). Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a history of interstitial lung disease.
* O2 saturation < 92% (on room air).
* Has unstable angina, new onset angina within the last 3 months, myocardial infarction within the last 6 months, and current congestive heart failure New York Heart Association Class III or higher. For Cohort 2: has ventricular arrhythmias, hypertensive urgency, or severe arterial thromboembolic events less than 6 months prior to study initiation.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the Screening visit through 120 days after the last dose of trial treatment. Women with a positive pregnancy test within 72 hours from Baseline.
* Has a positive Human immunodeficiency virus (HIV) positive test. Participants with HIV positive test on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Has known history of Chronic Hepatitis B or C. For participants with evidence of chronic hepatitis B virus (HBV) infection, if the HBV viral load is undetectable while on suppressive therapy the subject can participate on the study. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either MRI or computerized tomography (CT) scan, for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has received a live vaccine within 30 days of the planned start of study therapy. Seasonal flu vaccines or COVID-19 vaccines that do not contain live virus are permitted.
* Drainage of ascitic or pleural fluid 2 or more times in the 4 weeks prior to the first dose of study drug or permanent drain in place (eg, PleurX®) for ascites or pleural effusion symptom management.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of AGEN1423 or Botensilimab.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Every 8 weeks until EOT, for up to 2 years.
  The objective response rate (ORR) is defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria, using the modified intent-to-treat (mITT) analysis set

SECONDARY OUTCOMES:
Disease Control Rate | Every 8 weeks from first day of treatment until EOT for both cohorts up to 2 years.
  Disease control rate (DCR) defined as the sum of stable disease, partial and complete responses according to RECISTv1.1 criteria.
Median Duration of Overall Response (DOR) | Up to approximately 2 years
  Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per RECISTv1.1, until the first date that recurrent or progressive disease is objectively documented. Patients without progressive disease are censored at the date of last disease assessment.
Median Overall Survival (OS) | Up to 2 Years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Median Progression-free Survival | Every 8 weeks from first day of treatment until EOT for both cohorts up to 4 Years
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last dsease assessment.
Grade 3-5 Treatment-related Toxicity Rate | For Cohort 1 AE evaluated on Cycle 1 days 1 and 8, and Day 1 of each subsequent cycle (each cycle is 14 days). For Cohort 2 AE evaluated on Cycle 1 days 1, 8 and 15 of each cycle (each cycle is 28 days).
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Bockorny, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu